CLINICAL TRIAL: NCT00100451
Title: Aging, Exercise, and Hormonal Influences of Fat Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: ENDO-050-95S
Record Dates: First submitted 2004-12-30; First posted 2004-12-31 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Cardiovascular Disease
Keywords: Adipose tissue; Aging; Exercise; Lipolysis; Estrogens
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Exercise

INTERVENTIONS:
Procedure: exercise

SUMMARY:
The purpose of this study is to determine whether exercise alters the way in which the body stores and breaks down fat. A second objective is to evaluate how these effects are influenced by your age and gender. These studies are important because aging, male gender, and menopause are associated with an increased storage of abdominal fat which is frequently accompanied by diabetes, a high blood cholesterol level, high blood pressure and greater risks of heart attack, stroke, and death. Increasing evidence suggests that these abnormalities and many other effects of aging may be partly due to lack of exercise.

DETAILED DESCRIPTION:
The physiologic cause(s) of the age-related increase in total body and abdominal fat mass are not well-understood. The purpose of this study is to determine whether aging is associated with decreased whole body lipolytic and other metabolic responses to epinephrine and insulin, whether these responses may be augmented by exercise training or in older women by estrogen administration and to investigate whether such metabolic changes are related to reductions in abdominal adiposity. Our objectives in this project are as follows: (1) to characterize age and gender differences in lipolysis and other aspects of metabolism at rest and during graded dose epinephrine infusion with or without a pancreatic islet clamp in healthy non-obese men and women aged 20-40 and 55-75 years, (2) to evaluate relationships between metabolic responses to epinephrine or insulin and portally and nonportally-drained visceral and subcutaneous adipose tissue mass in these individuals, (3) to delineate the effects of acute and chronic exercise on lipolytic and other metabolic responses to epinephrine and insulin and on adipose tissue distribution in healthy younger and older men and women, and (4) to investigate whether 7 days and 12 months or estrogen and cyclic progesterone replacement therapy or placebo in healthy 55-75 year old women alter lipolytic and other metabolic responses to epinephrine and insulin and adipose tissue distribution.

The rates of lipolysis, oxygen uptake, fat and carbohydrate oxidation, and total triglyceride-free fatty acid (FFA) substrate cycling will be determined by indirect calorimetry and by gas chromatography-mass spectrometric analyses of blood samples obtained during infusions of the stable isotope tracers [D5] glycerol and [1 -13C] palmitate in the baseline state, during a pancreatic islet clamp in half of all male and female participants, and in all participants during a subsequent 4-stage graded dose epinephrine infusion. These data will be expressed in relation to total body wieght, fat mass, and fat-free mass, assessed from measurements of body density made by hydrostatic weighing. Adipose tissue distribution will be characterized by determination of the cross-sectional area and volume of portally and nonportally-drained visceral and subcutaneous fat deposits identified by radiographic density criteria on computed tomographic scans obtained at the level of the nipple, umbilicus, gluteal region, and midthigh. Insulin action on glucose disposal will be assessed during a hyperinsulinemic euglycemic clamp. Age and gender differences and their interactions with exercise and the plasma epinephrine concentration in the baseline state and during submaximally and maximally stimulating rates of epinephrine infustion will be evaluated by analysis of variance and covariance. Relationships between effects of estrogen treatment or exercise of adipose tissue distribution and responses to epinephrine and insulin will be assessed by multiple regression analysis.

We hypothesize that increased age will be associated with lower epinephrine-induced rates of lipolysis, fat oxidation, and triglyceride-FFA substrate cycling and decreased insulin action in both men and women when expressed in relation to total fat mass. We further hypothesize that these age-related differences will be at least partly ameliorated by exercise training and by treatment with estrogen in conjunction with a decrease in visceral abdominal and total body adiposity.

ELIGIBILITY:
* Healthy men or women between the ages of 20 and 75

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1994-06; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Locations (1):
- VA Medical Center, St Louis, Missouri, United States